CLINICAL TRIAL: NCT05667493
Title: An Open-Label Extension Study to Assess the Long-Term Safety of Eplontersen (ION-682884) in Patients With Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR-CM)
Brief Title: An Extension Study to Assess Long-Term Safety of Eplontersen in Adults With Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR-CM)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ION-682884-CS12; 2022-000826-74 (EudraCT Number)
Record Dates: First submitted 2022-07-12; First posted 2022-12-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR CM)
Keywords: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — eplontersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eplontersen (Experimental): Eplontersen will be administered once every month by sub-cutaneous (SC) injection for up to 36 months or 6 months after eplontersen is approved and available in the site's country, whichever occurs first.
  Interventions: Drug: Eplontersen

INTERVENTIONS:
Drug: Eplontersen — Eplontersen will be administered by SC injection.
  Other Names: ION-682884; IONIS-TTR-LRx

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of extended dosing with eplontersen in participants with ATTR-CM.

DETAILED DESCRIPTION:
This is a multicenter, open-label extension, Phase 3 study in up to approximately 1400 participants from the 682884-CS2 study. Eligible participants will receive eplontersen once every 4 weeks for up to 36 months or until after eplontersen is approved and available in the site's country, whichever occurs first. Participants will also receive daily supplemental doses of the recommended daily allowance (RDA) of vitamin A.

ELIGIBILITY:
Inclusion Criteria:

1. Satisfactory completion of Treatment Period and the End of Treatment Visit of the Index Study (ION-682884-CS2) OR diagnosis of ATTR-CM and satisfactory participation on ISIS 420915- CS101 study as judged by the Investigator and Sponsor.
2. Investigator is willing to treat the participant with open-label eplontersen.
3. Willingness to adhere to vitamin A supplementation per protocol.

Exclusion Criteria:

1. Permanently discontinued study drug administration while participating in the Index Study (ION 682884-CS2) or IST (ISIS 420915-CS101 Study).
2. Have any new condition or worsening of an existing condition that in the opinion of the Investigator or Sponsor would make the participant unsuitable for enrolment, or which could interfere with the participant participating in or completing the study, including the need for treatment with medications disallowed in the Index Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) | Baseline up to 36 months
Change From Baseline in Platelet Count | Baseline up to 36 months
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline up to 36 months
Change From Baseline in Urine Protein Creatinine Ratio (UPCR) | Baseline up to 36 months

SECONDARY OUTCOMES:
Change From Baseline in Transthyretin (TTR) Serum Levels | Baseline up to 36 months
Change From Baseline in 6-minute Walk Test (6MWT) | Baseline up to 36 months
Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline up to 36 months

CONTACTS AND LOCATIONS:
Locations (122):
- United States (46):
  - Mayo Clinic, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Altman Clinical and Translational Research Institute - Center for Clinical Research, La Jolla, California
  - University Of California San Francisco Urology Practice, San Francisco, California
  - Stanford University (Leland Stanford Junior University), Stanford, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The George Washington Medical Faculty Associates - Foggy Bottom North Pavilion, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Heart of Fayetteville, Atlanta, Georgia
  - Emory Heart and Vascular Center - Emory Clifton Campus, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Fayetteville, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Allina Health Minneapolis Heart Institute - Abbott Northwestern's Heart Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - New York University Langone Cardiology Associates, New York, New York
  - Weill Cornell Medicine Cardiology, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carl and Edyth Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Heart and Vascular Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires
- Australia (9):
  - Advara HeartCare, Joondalup, Western Australia
  - Advara HeartCare Murdoch, Murdoch, Western Australia
  - Box Hill Hospital, Clayton
  - Royal Hobart Hospital, Hobart
  - Advara HeartCare - Joondalup, Joondalup
  - Liverpool Hospital, Liverpool
  - Advara HeartCare Murdoch, Murdoch
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Limbourg
- Brazil (7):
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - A Beneficência Portuguesa de São Paulo - Unidade Mirante, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coração de São Paulo, São Paulo
  - Universidade Estadual de Campinas, São Paulo
  - Centro Avançado de Pesquisa e Estudos para o Diagnóstico CAPED, São Paulo
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital Regional de Rimouski, Rimouski
  - Gordon and Leslie Diamond Health Care Centre, Vancouver
- Czechia (3):
  - Fakultní Nemocnice u sv. Anny v Brně, Brno
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Institut Klinické a Experimentální Medicíny, Prague
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hôpital de la Timone, Marseille
  - Centre Hospitalier Universitaire De Nantes - Hôpital Nord Laennec, Nantes
  - Hôpital Haut-Lévêque, Pessac
  - Hôpital Rangueil, Toulouse
- Germany (5):
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Heidelberg - Zentrum für Innere Medizin, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Würzburg
- General Hospital of Athens "Alexandra", Athens, Greece
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
- Italy (6):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedale Università di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanita Pubblica, Pisa
  - Azienda Ospedaliera - Universitaria Sant' Andrea, Roma
- Japan (3):
  - Kurume University Hospital, Kurume-Shi, Fukuoka
  - Saiseikai Fukuoka General Hospital, Fukuoka, Hukuoka [Fukuoka]
  - Kumamoto University Hospital, Kumamoto
- Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow, Poland
- Portugal (7):
  - Hospital da Senhora da Oliveira, Guimarães
  - Unidade Local de Saúde do Alto Ave, E. P. E (Hospital da Senhora da Oliveira Guimarães), Guimarães
  - Unidade Local de Saúde de São José, E. P. E - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar Universitário do Porto - Hospital Geral de Santo Antonio, Porto
  - Unidade Local de Saúde de Santo António, E. P. E - Hospital Geral de Santo Antonio, Porto
  - Centro Hospitalar Universitário de São João, Porto
  - Unidade Local de Saúde de São João, EPE, Porto
- Spain (4):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skellefteå lasarett, Skellefteå
- United Kingdom (6):
  - AES - Synexus - Scotland Clinical Research Centre, Bellshill, England
  - AES - Synexus - Midlands, Edgbaston, England
  - Synexus - Manchester Clinical Research Centre, Manchester, England
  - AES - Synexus - Wales, Cardiff, Wales
  - Royal Free London NHS Foundation Trust, Hampstead
  - Richmond Pharmacology, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.